CLINICAL TRIAL: NCT03716596
Title: Study on the Safety and Therapeutic Effect of Stereotactic Body Radiotherapy and Anti-PD-1 Antibody in Late Stage or Recurrent Pancreatic Cancer Patients Who Failed in Second-line Chemotherapy
Brief Title: SBRT and Anti-programmed Cell Death Protein 1(Anti-PD-1) in Late Stage or Recurrent Pancreatic Cancer Patients
Acronym: CISPD-2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The effect of the regime was not satisfied
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISPD-2
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; Second-line Chemotherapy resistant; immune therapy; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; spartalizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT and PD-1 (Experimental): Stereotactic body radiotherapy, radiation dose is 40-50 Gy in total. Intravenous drug of anti-PD-1 antibody, 200mg, once a time, every three weeks.
  Interventions: Radiation: SBRT; Drug: anti-PD-1 antibody

INTERVENTIONS:
Radiation: SBRT — SBRT radiation dose is 40-50 Gy in total.
  Other Names: Stereotactic Body Radiotherapy
Drug: anti-PD-1 antibody — Intravenous drug of anti-PD-1 antibody, 200mg, once a time, every three weeks.
  Other Names: keytruda

SUMMARY:
When gemcitabine based chemo and fluorouracil based chemo regimes are failed in late-stage or recurrent pancreatic cancer patients, there is no alternative options. Anti-PD-1 antibody has became a promising anti-cancer drug. While it showed limited efficacy in pancreatic cancer. Stereotactic Body Radiotherapy has been a new method to locally treat metastatic cancer. This study is aimed to evaluate the safety and efficacy of the combination of SBRT and anti-PD-1 antibody in late-stage or recurrent pancreatic caner who failed in second-line chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer is a kind of cancer with poor prognosis. Nowadays, recommended treatment for late-stage or recurrent pancreatic cancer patients are fluorouracil based chemotherapy (such as FOLFIRINOX) and gemcitabine based chemotherapy. When these two chemo regimes are failed, however, there is no alternative options. With the improvement of immune therapy, anti-PD-1 antibody has became a promising anti-cancer drug. While it showed limited efficacy in pancreatic cancer. Stereotactic Body Radiotherapy (SBRT) has been a new method to locally treat metastatic cancer. And previous studies showed that SBRT may enhance the efficacy of immunotherapy. So this study is amed to evaluate the safety and efficacy of the combination of SBRT and anti-PD-1 antibody in late-stage or recurrent pancreatic caner who failed in second-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.≥18 years.
* 2.Histopathology or cytology confirmed pancreatic cancer.
* 3.Patients failed in second-line chemotherapy: patients have failed in gemcitabine-based chemotherapy and also failed in fluorouracil-based chemotherapy (like FOLFIRINOX), failed in combination of chemotherapy and radiotherapy; patients may have failed in immune therapy (including anti-PD-1 antibody).
* 4. Eastern cooperative oncology group physical fitness score was 0~2.
* 5. The main organs are functional and meet the following criteria (Routine blood tests were in accordance with the following criteria):

  1. White blood cell (WBC) ≥3.5 x 10^6 /L, neutrophil >1.5 x10^9/L,
  2. platelet (PLT) ≥50 x10^9/L,
  3. hemoglobin (HB) ≥80 g/L,
  4. total bilirubin (TB) ≤1.5 x ULN (upper limit of normal value). 5）Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2 x ULN (upper limit of normal value) (if there is liver metastasis, ≤ 5 x ULN).

  6) Serum creatinine (Scr) ≤ 1.5 x ULN 7) Albumin (ALB) ≥ 3 g/dL.
* 6. Patients will be informed consent, and understand and are willing to cooperate with the trial and sign related documents.

Exclusion Criteria:

* 1. In the first 4 weeks before the start of the study, they took part in other drug clinical trials.
* 2. Before the start of the study, they were diagnosed as immune deficiency diseases or need systemic steroid therapy.
* 3. In the first 4 weeks before the start of the study, they took anti-tumor immune therapy; or didn't recovery from the adverse effects caused by the anti-tumor immune therapy.
* 4. In the first 2 weeks before the start of the study, they took chemotherapy, small molecule targeting therapy, and radiotherapy; or didn't recovery from the adverse effects caused by these therapies.
* 5. Has had active tuberculosis before.
* 6. Has a history of malignant tumor, except for basal and skin squamous cell carcinoma, cervical carcinoma in situ and papillary thyroid carcinoma.
* 7. Has central nervous system metastasis or meningeal metastasis.
* 8. Has serious and uncontrollable internal diseases such as severe diabetes, severe hypertension, serious infection, congestive heart failure, ventricular fibrillation, coronary heart disease with obvious symptoms or myocardial infarction in the past 6 months.
* 9. Has blood precancerous diseases, such as myelodysplastic syndrome.
* 10. Has clinically relevant or preexisting interstitial lung diseases, such as noncommunicable pneumonia or pulmonary fibrosis, or evidence of interstitial lung diseases on baseline chest CT scans or chest x-rays.
* 11. Past or physical examinations have found diseases of the central nervous system, with the exception of those that have been adequately treated (such as primary brain tumors, uncontrolled seizures or strokes with standard medication).
* 12. Has preexisting neuropathy at > level 1 (NCI CTCAE).
* 13. Allotransplantation requires immunosuppression therapy or other major immunosuppression therapy.
* 14. Has a severe open wound, ulcer, or fracture.
* 15. Systemic treatment is required for autoimmune diseases that have been active for the past 2 years.Alternative therapies are not systemic treatments.
* 16. Has a history of non-infectious pneumonia requiring steroid therapy or active pneumonia.Has interstitial lung disease.
* 17. Patients with active infections require systemic treatment.
* 18. Patients with active hepatitis b or c are not included in liver lesions SBRT.
* 19. Has vaccinate within 30 days before treatment.Including intranasal influenza vaccines, except seasonal influenza vaccines
* 20. Others: allergic history of similar drugs, pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to approximately 12 months
  The percentage of people still alive for a given period of time after diagnosis

SECONDARY OUTCOMES:
Disease control rate | Up to approximately 12 months
  Percentage of patients whose cancer doesn't progress after treatment
Objective response rate | Up to approximately 12 months
  Percentage of patients whose cancer shrinks or disappears after treatment
Progression-free survival | Up to approximately 12 months
  The percentage of people does not get worse for a period of time after diagnosis
EORTC quality of life questionnaire (QLQ) | Up to approximately 12 months
  Assessed by the European Organization for Research and Treatment of Cancer Quality of Life
Common Toxicity Criteria for Adverse Effects | Up to approximately 12 months
  According to Common Toxicity Criteria for Adverse Effects version 4
Related tumor markers | Up to approximately 12 months
  Serum level of related tumor markers (like carbohydrate antigen19-9, carcinoembryonic antigen and so on)

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, MD PhD, Principal Investigator — second affiliated hospital, Zhejiang University School of Medicine
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided